CLINICAL TRIAL: NCT00722579
Title: A Non-Randomized, Multi-Center, Single-Arm Safety Study of the Presillion Stent in de Novo Native Coronary Artery Lesions
Brief Title: A Study of the Presillion Stent in de Novo Coronary Lesions
Acronym: PRESILLION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Hans-Peter Stoll, MD, Cordis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC08-01
Record Dates: First submitted 2008-07-24; First posted 2008-07-25 (Estimated); Last update posted 2010-06-14 (Estimated); Status verified 2010-06

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): The PRESILLION TM Coronary Stent is an L-605 cobalt chromium (CoCr) stent.
  Interventions: Device: PRESILLION cobalt chromium stent

INTERVENTIONS:
Device: PRESILLION cobalt chromium stent — PTCA with bare-metal stent
  Other Names: bare-metal stent

SUMMARY:
The PRESILLION Study is a non-randomized, multi-center, single-arm study evaluating the safety of an approved Cobalt Chromium bare metal stent system for the treatment of ischemic heart disease attributable to a stenotic de novo lesion in a native coronary artery.

The study population will include 100 patients with up to two de novo native coronary artery lesions with a maximum lesion length of 30mm in a maximum of two major coronary arteries with reference vessel diameter >= 2.5mm and <= 4.0mm by visual estimation. Patients will be followed for 1 month and 6 month post-procedure for assessment of MACE and all other adverse events.

DETAILED DESCRIPTION:
The PRESILLION Stent System is intended for use in patients with symptomatic ischemic heart disease attributable to stenotic de novo lesions of native coronary arteries with reference vessel diameter from 2.5 mm to 4.0 mm with a lesion length up to 30 mm that are amenable to percutaneous treatment with coronary stenting. The stent is intended as a permanent implanted device.

The primary objective of this study is to evaluate the safety of the PRESILLION Stent System in the treatment of de novo stenotic lesions in native coronary arteries. The primary safety measure is the composite of MACE up to one (1) month follow up. The MACE rate shall meet the performance goal for bare metal stents in order to show the safety of the device.

The protocol has been amended and data will be collected for a time point as close as possible to (but after) the 6 months post index procedure in a non-interventional and retrospective manner. The data point will contain exactly the same follow-up information as was collected during the 1 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be >= 18 years of age.
* Patient is eligible for percutaneous coronary intervention (PCI).
* Acceptable candidate for coronary artery bypass surgery (CABG).
* Female patients of childbearing potential must have a negative pregnancy test within 7 days prior to enrolment and utilize reliable birth control for trial duration.
* Diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS I, II, III, IV) or unstable angina pectoris (Braunwald Classification B&C, I-II-III) or patients with documented silent ischemia.
* Treatment of up to two de novo native coronary artery lesions in a maximum of two major coronary arteries.
* Target reference vessel diameter of both lesions must be >= 2.5mm and <= 4.0mm in diameter (visual estimate).
* Target lesion length must be <= 30mm and be covered by one study stent.
* Target lesion stenosis for both lesions is > 50% and < 100% (visual estimate).
* At least TIMI I coronary flow.
* Patient is willing to comply with the specified follow-up evaluation.
* Patient must provide written informed consent prior to the procedure using a form that is approved by the local Ethics Committee.

Exclusion Criteria:

* Recent myocardial infarction (either STEMI or non STEMI < 48 hours prior to planned index procedure).
* The patient has unstable angina classified as Braunwald A I-II-III.
* The patient has unprotected left main coronary artery disease (stenosis >50%).
* A significant (> 50%) stenosis proximal or distal to the target lesion.
* Angiographic evidence of thrombus within the target lesion.
* Heavily calcified lesion and/or calcified lesion, which cannot be successfully predilated and/or an excessively tortuous vessel which makes it unsuitable for stent delivery and deployment.
* Left ventricular ejection fraction <= 25%.
* Totally occluded lesion (TIMI 0 level).
* The patient has impaired renal function (creatinine 3.0mg/dL) at the time of treatment.
* The patient had a Cerebrovascular Accident (CVA) within the past 6 months.
* Prior stent within 10mm of target lesion.
* The target lesion is ostial in location (within 3.0mm of vessel origin).
* The target lesion involves a bifurcation with a diseased (>50% stenotic) branch vessel >= 2.0mm in diameter (or side branch requiring intervention of protection).
* The target lesion is located in a bypass graft. Note: stenting of lesions in bypassed native coronary arteries is allowed.
* Known allergies to the following: aspirin, clopidogrel bisulfate (Plavix ®) and ticlopidine (Ticlid ®), heparin, cobalt chromium, contrast agent (that cannot be managed medically).
* The patient has any significant medical condition which in the investigator's opinion may interfere with the patient's optimal participation in the study.
* The patient is currently participating in an investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the study endpoints.
* Intervention of another lesion within 30 days prior to, or is planned or highly probably to be performed 30 days after the index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2008-07; Primary Completion 2008-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Composite of MACE which includes cardiac death, myocardial infarction (Q-wave and non Q-wave) and clinically driven target lesion revascularization (TLR). | 1-month and 6-months post-procedure

SECONDARY OUTCOMES:
Clinically driven Target Lesion Revascularization (TLR) defined as repeat PCI or CABG to the target lesion. | 1-month and 6-months post-procedure
Clinically driven Target Vessel Revascularization (TVR) defined as repeat PCI or CABG to the target vessel. | 1-month and 6-months post-procedure
Target Vessel Failure (TVF) defined as target vessel revascularization, recurrent myocardial infarction, or cardiac death that could not be clearly attributed to a vessel other than the target vessel. | 1-month and 6-months post-procedure
Myocardial Infarction (MI). | 1-month and 6-months post-procedure
Major bleeding. | 1-month and 6-months post-procedure
Device success. | Post-procedure
Lesion success. | Post-procedure
Procedure success. | Post-procedure
Incidence of acute and sub-acute stent thrombosis according the ARC definition. | 1-month and 6-months post-procedure
Stroke. | Post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: V. Legrand, MD, Phd, Principal Investigator — Centre Hospitalier Universitaire de Liege
Locations (1):
- CHU de Liège, Liège, Belgium